CLINICAL TRIAL: NCT01071668
Title: Feasibility Study to Develop the Analysis of the Metabolome During the Onset of Labor During Pregnancy
Brief Title: Onset of Labor and Metabolomics (GEM-2)
Acronym: GEM-2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, Dr, Université de Sherbrooke
Other Study IDs: 09-041
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Pregnancy
Keywords: onset of labor; metabolomics; vaginal secretions; urine; blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal secretions, whole blood and urine are collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GEM-2 Cohort: Women who have a low risk pregnancy before onset of labor. Patients included in the study who will be hospitalized with spontaneous labor at term with intact membranes or preterm labor will be included in the study group. Patients with premature rupture of membranes or induction of labor will be analyzed separately.

SUMMARY:
Premature birth is a public health problem and its incidence has recently increased in all developed countries. In Canada, it represented 6.4% of births in 1981 and 7.6% in 2000. In the last decade, the survival rate of premature infants has increased considerably, but neurological vulnerability has not changed. Premature births are the cause of approximately 28% of neonatal mortality in the world and is the major cause of perinatal mortality and morbidity in developed countries.

Approximately 75-80% of preterm births are spontaneous preterm birth. This type of premature birth included the preterm labor and premature rupture of membranes before term. The contractile activity represents one of the fundamental properties of the uterus during pregnancy and childbirth. The abnormalities associated with uterine contractions are the cause of pathological conditions with important consequences for the mother and fetus.

Metabolomics involves a new technology to investigate small molecules that characterize biochemical pathways of interest. The change in concentration levels of these molecules in various biological samples such as urine and blood in the presence of a disease or a patient can be particularly useful for identifying new biomarkers.

The hypothesis of this study is that gestational metabolomes detected in maternal fluids differ according to pathological situations and lead to the initiation of spontaneous labor. The whole research program has two complementary objectives in order to expect a decrease of prematurity: a) better understanding of all the physiological mechanisms leading to prematurity and b) better identification of patients at high risk for a better management of these women.

DETAILED DESCRIPTION:
Metabolomics involves a new technology using the methods of separation and detection complex to investigate a set of small molecules that characterize biochemical pathways of interest. The change in concentration levels of these molecules in various biological samples such as urine and blood in the presence of a disease or a patient can detect metabolic fingerprints that can be particularly useful for identifying new biomarkers. These will thereafter be quantified and validated by metabolic profiling. To our knowledge, there are few studies on metabolomics and pregnancy.

Methods:

The studied population will be pregnant women between 20-30 weeks of gestation without any obstetrical complications.

Vaginal secretions, blood and urine samples will be taken:

* After inclusion in the project
* At hospital admission for delivery
* During labor

Blood and urine sample will also be taken:

* 48 hours after delivery
* 6-8 weeks after delivery

ELIGIBILITY:
Inclusion Criteria:

* Women with single pregnancy
* Adults (> 18 years old)

Exclusion Criteria:

* Women with a severe congenital fetal malformation
* Fetal death
* Preexisting hypertension (ie before 20 weeks of gestation)
* Anti-phospholipid syndrome
* Lupus,
* Nephropathy, etc.
* Viral infections (HIV or hepatitis)
* Women who want an elective Caesarean section are excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women between 20-30 weeks of gestation who have a low risk pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
comparison between the metabolic patterns of women before and during labor | one and half year

SECONDARY OUTCOMES:
The study also looks at the comparison of metabolic patterns in late pregnancy and postpartum. | one and half year
The project will characterize the metabolome in different fluids collected | one and half year
The study will compare the metabolome of women with spontaneous onset of labor with that of women with premature rupture of membranes or induction of labor | one and half year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Centre Hospitalier de l'Université de Sherbrooke
Locations (1):
- Centre Hospitalier de l'Université de Sherbrooke, Sherbrooke, Quebec, Canada